CLINICAL TRIAL: NCT00538707
Title: Effect of Mental Stress on Platelet Function in Healthy Subjects
Brief Title: Effect of Mental Stress on Platelet Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: University of Zurich, University Hospital Zurich
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EK-1382
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Mental Stress
Keywords: mental stress; platelet adhesion; platelet function; catecholamines
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young subjects (Experimental)
  Interventions: Behavioral: 2-minute Bondet test
- Older subjects (Experimental)
  Interventions: Behavioral: 2-minute Bondet test

INTERVENTIONS:
Behavioral: 2-minute Bondet test — 2-minute Bondet test
  Other Names: 2-minute Bondet light test

SUMMARY:
The aim of the project is to study the acute and chronic effect of mental stress on platelet adhesion and aggregation in two population composed of normal subjects at different ages

DETAILED DESCRIPTION:
Psychological stress is an important cardiovascular risk factor. Activation of platelets plays an important role in atherosclerosis development and it could be one of the mechanisms linking psychological stress and cardiovascular diseases.

We plan to include 32 healthy subjects. (16 in every group). One group with subjects at age 20 - 49 and the other group with subjects at age 50 - 70 years.

The aim of the study will be to assess the acute and chronic effect of a standard short mental stress (2-minute Bondet Test) on platelet function and of the level of endothelin-1, catecholamines and cortisol. We plan to evaluate if age may play a role in the effect of psychological stress on platelet function.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects between 20 - 70 years of age
* written informed consent
* no evidence of diseases

Exclusion Criteria:

* pregnancy
* oral contraceptives
* smoking
* use of aspirin or NSAIDs within the last week
* use of benzodiazepines within the last week
* Alcohol or drug abuse
* participation in another study within the last month

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of platelet function (shear stress dependent platelet adhesion and aggregation) before and after mental stress | 60 minutes

SECONDARY OUTCOMES:
Evaluation of the plasma level of endothelin, catecholamines and salivary cortisol level before and after mental stress | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Georg Noll, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland